CLINICAL TRIAL: NCT05959525
Title: Correlation Between the Dental Arch Morphology and the Articular Eminence Height and Inclination on CBCT Scans of an Egyptian Population: A Cross-Sectional Study.
Brief Title: Correlation Between Dental Arch and Articular Eminence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Mohamed Khaled Hassan Mohamed Ali, Dr. Sarah Khaled, Cairo University
Other Study IDs: Dental arch&Articular eminence
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Articular Eminence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ovoid dental arch
- Square dental arch
- Tapered dental arch

SUMMARY:
the aim of the study is to assess the correlation between the dental arch morphology and the articular eminence height and inclination by using CBCT scans of a sample of the Egyptian population.

ELIGIBILITY:
Inclusion Criteria:

* • CBCT scans of adult Egyptian patients, males and females with ages starting from 18 till 45.

  * Scans of patients who have complete set of permanent dentitions (third molars are not considered), or at least not more than one tooth is missed in each arch.
  * CBCT scans with field of view that shows the full view of TMJ.

Exclusion Criteria:

* • CBCT scans of patients with fractures in the articular bone surfaces.

  * CBCT scans of patients with pathological lesions in the TMJ or articular eminence.
  * CBCT scans with artifacts that could interfere with the assessment of the articular eminence and dental arches.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: A group of dentated Egyptian people
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between the morphology of the dental arch and the articular eminence inclination. | Baseline

SECONDARY OUTCOMES:
Correlation between the morphology of the dental arch and the articular eminence height. | Baseline
Correlation between the dental arch measurements and the articular eminence height and inclination measurements. | Baseline

REFERENCES:
- [Background] Bertram F, Hupp L, Schnabl D, Rudisch A, Emshoff R. Association Between Missing Posterior Teeth and Occurrence of Temporomandibular Joint Condylar Erosion: A Cone Beam Computed Tomography Study. Int J Prosthodont. 2018 January/February;31(1):9-14. doi: 10.11607/ijp.5111. Epub 2017 Nov 16. PMID 29145525
- [Background] Costa EDD, Peyneau PD, Roque-Torres GD, Freitas DQ, Ramirez-Sotelo LR, Ambrosano GMB, Verner FS. The relationship of articular eminence and mandibular fossa morphology to facial profile and gender determined by cone beam computed tomography. Oral Surg Oral Med Oral Pathol Oral Radiol. 2019 Dec;128(6):660-666. doi: 10.1016/j.oooo.2019.07.007. Epub 2019 Jul 18. PMID 31494114
- [Background] Dzingute A, Pileicikiene G, Baltrusaityte A, Skirbutis G. Evaluation of the relationship between the occlusion parameters and symptoms of the temporomandibular joint disorder. Acta Med Litu. 2017;24(3):167-175. doi: 10.6001/actamedica.v24i3.3551. PMID 29217971
- [Background] Fan XC, Ma LS, Chen L, Singh D, Rausch-Fan X, Huang XF. Temporomandibular Joint Osseous Morphology of Class I and Class II Malocclusions in the Normal Skeletal Pattern: A Cone-Beam Computed Tomography Study. Diagnostics (Basel). 2021 Mar 18;11(3):541. doi: 10.3390/diagnostics11030541. PMID 33803644
- [Background] Hamza MK, Shantha AM, Ashwathappa DT, Rajanna S, Puttegowda AK. Assessing the Articular Eminence Asymmetry in Dentate, Partially Edentulous and Edentulous patients Using Cone-Beam Ct. J Pharm Bioallied Sci. 2021 Jun;13(Suppl 1):S667-S671. doi: 10.4103/jpbs.JPBS_685_20. Epub 2021 Jun 5. PMID 34447177
- [Background] Hou X, Xu X, Zhao M, Kong J, Wang M, Lee ES, Jia Q, Jiang HB. An overview of three-dimensional imaging devices in dentistry. J Esthet Restor Dent. 2022 Dec;34(8):1179-1196. doi: 10.1111/jerd.12955. Epub 2022 Aug 15. PMID 35968802
- [Background] Ilguy D, Ilguy M, Fisekcioglu E, Dolekoglu S, Ersan N. Articular eminence inclination, height, and condyle morphology on cone beam computed tomography. ScientificWorldJournal. 2014 Feb 13;2014:761714. doi: 10.1155/2014/761714. eCollection 2014. PMID 24696193
- [Background] Matsuda S, Yamaguchi T, Mikami S, Yoshimura H, Gotouda A. Can malocclusion provide clinicians with information for differential diagnosis of temporomandibular joint diseases?: A review. Medicine (Baltimore). 2022 Aug 19;101(33):e29247. doi: 10.1097/MD.0000000000029247. PMID 35984194
- [Background] Moscagiuri F, Caroccia F, Lopes C, Di Carlo B, Di Maria E, Festa F, D'Attilio M. Evaluation of Articular Eminence Inclination in Normo-Divergent Subjects with Different Skeletal Classes through CBCT. Int J Environ Res Public Health. 2021 Jun 3;18(11):5992. doi: 10.3390/ijerph18115992. PMID 34204929
- [Background] Othman SA, Xinwei ES, Lim SY, Jamaludin M, Mohamed NH, Yusof ZY, Shoaib LA, Nik Hussein NN. Comparison of arch form between ethnic Malays and Malaysian Aborigines in Peninsular Malaysia. Korean J Orthod. 2012 Feb;42(1):47-54. doi: 10.4041/kjod.2012.42.1.47. Epub 2012 Feb 27. PMID 23112931
- [Background] Omar H, Alhajrasi M, Felemban N, Hassan A. Dental arch dimensions, form and tooth size ratio among a Saudi sample. Saudi Med J. 2018 Jan;39(1):86-91. doi: 10.15537/smj.2018.1.21035. PMID 29332114
- [Background] Reissmann DR, Anderson GC, Heydecke G, Schiffman EL. Effect of Shortened Dental Arch on Temporomandibular Joint Intra-articular Disorders. J Oral Facial Pain Headache. 2018 Summer;32(3):329-337. doi: 10.11607/ofph.1910. PMID 30036887
- [Background] Sumbullu MA, Caglayan F, Akgul HM, Yilmaz AB. Radiological examination of the articular eminence morphology using cone beam CT. Dentomaxillofac Radiol. 2012 Mar;41(3):234-40. doi: 10.1259/dmfr/24780643. Epub 2011 Nov 10. PMID 22074873
- [Background] Verner FS, Roque-Torres GD, Ramirez-Sotello LR, Devito KL, Almeida SM. Analysis of the correlation between dental arch and articular eminence morphology: a cone beam computed tomography study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2017 Oct;124(4):420-431. doi: 10.1016/j.oooo.2017.07.004. Epub 2017 Jul 26. PMID 28847629
- [Background] Virlan MJR, Paun DL, Bordea EN, Pellegrini A, Spinu AD, Ivascu RV, Nimigean V, Nimigean VR. Factors influencing the articular eminence of the temporomandibular joint (Review). Exp Ther Med. 2021 Oct;22(4):1084. doi: 10.3892/etm.2021.10518. Epub 2021 Jul 30. PMID 34447477
- [Background] Zhang J, Jiao K, Zhang M, Zhou T, Liu XD, Yu SB, Lu L, Jing L, Yang T, Zhang Y, Chen D, Wang MQ. Occlusal effects on longitudinal bone alterations of the temporomandibular joint. J Dent Res. 2013 Mar;92(3):253-9. doi: 10.1177/0022034512473482. Epub 2013 Jan 22. PMID 23340211